CLINICAL TRIAL: NCT02684084
Title: Combination OZURDEX® & LUCENTIS® vs. OZURDEX® Monotherapy in Incomplete-Responders With Diabetic Macular Edema: The COLLIDE Trial
Brief Title: Combination OZURDEX® & LUCENTIS® vs. OZURDEX® Monotherapy in Incomplete-Responders With Diabetic Macular Edema
Acronym: COLLIDE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study revised significantly. New trial to be launched.
Sponsor: North Toronto Eye Care Laser and Eye Specialists (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Pradeepa Yoganathan, Principal Investigator, North Toronto Eye Care Laser and Eye Specialists
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT-CAN-EYE-0399
Record Dates: First submitted 2015-11-26; First posted 2016-02-17 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic Macular Edema; Ozurdex; Lucentis
MeSH Terms: interventions — Calcium Dobesilate; Dexamethasone; Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combination group (RBZ+DEX) (Active Comparator): 30 eyes will receive an intravitreal Lucentis (0.5 mg) injection followed by Ozurdex implant (0.7 mg) injection within 0 to 8 days.
  Interventions: Drug: Ozurdex; Drug: Lucentis
- Monotherapy group (DEX only) (Active Comparator): 30 eyes will receive Ozurdex implant (0.7 mg) injection only
  Interventions: Drug: Ozurdex

INTERVENTIONS:
Drug: Ozurdex — OZURDEX® (DEX implant; Allergan Inc. Irvine, CA, USA) is a sustained-release biodegradable implant approved for treatment of Macular Edema secondary to central retinal vein occlusion as well as noninfectious uveitis affecting the posterior segment
  Other Names: DEX implant, dexamethasone
Drug: Lucentis — LUCENTIS® (0.5 mg ranibizumab or RBZ, an anti-neovascular VEGF-A inhibitor, Novartis Pharmaceuticals Canada Inc.) was the first approved medical treatment for DME
  Other Names: Ranibizumab
  Arms: Combination group (RBZ+DEX)

SUMMARY:
This is a 24-week, prospective, multi-center, open-label, randomized, investigator-initiated pilot study to explore the effects of RBZ (0.5 mg) plus DEX implant (0.7 mg) PRN combination therapy (n = 30) vs. DEX implant PRN monotherapy (n = 30) in pseudophakic eyes with center-involved DME that have demonstrated prior incomplete response to 3-6 anti-VEGF treatments.

DETAILED DESCRIPTION:
1. Hypothesis

   Pseudophakic center-involved DME eyes with incomplete response to 3-6 anti-VEGF injections (i.e., RBZ, BCZ or IAI) will have similar visual acuity gains, as assessed with AUC analysis (change from baseline randomization (Time 0) BCVA letters through 24 weeks ± 1 week), with a combination treatment regimen consisting of RBZ (0.5 mg) and DEX implant (0.7 mg) vs. a monotherapy treatment regimen with DEX implant (0.7 mg).
2. Description of Study procedures:

   Screening (Visit 1): At this initial visit, the study doctor or delegate will explain the study to the patient, answer all of their questions, and will ask them to sign an informed consent form. If the patient agrees to participate in the study, the study doctor or delegate will perform routine examinations; ask them questions about their past medical history, current medical conditions, and all medication or treatments they are receiving. If the patient is female, they may have a urine pregnancy test performed. Patients will undergo your regular eye evaluations. If their glycosylated hemoglobin (HbA1a) level is not available within 12-15 weeks of Visit 1 an HbA1c test will be performed at screening. Patients will be assigned to one of two possible treatment regimens (1.) combination consists of LUCENTIS® (0.5 mg) followed by OZURDEX® (0.7 mg) 0-8 days later or (2.) OZURDEX® (0.7 mg) monotherapy. This visit will last approximately 1-2 hours. Patients will always have the choice of receiving both medications at the same time or split between 2 shorter visits.

   Baseline/Randomization (Visit 2): If patients are eligible to receive study treatment(s) they will be scheduled for a baseline randomization study visit to allow collection of eye exam data (intraocular pressure, inflammatory cells, abnormal blood vessels) and ocular coherence tomography OCT. This is the same type of eye exam and OCT patients typically undergo at a retina specialist's office. Additionally, patients will undergo a special vision test and an intravenous fluorescein angiogram to assess retinal circulation. This visit will last approximately 2 hours. The next study visit (Visit 3) will be scheduled in 4-5 weeks. Someone from your study doctor's office will contact the patient prior to the baseline visit to remind you of this next visit

   Week 4 (Visit 3): This study visit will allow collection of eye exam data, vision, eye pressure, and OCT. This visit will last approximately 1 hour. The next study visit (Visit 4) will be scheduled in 4-5 weeks. Someone from the study doctor's office will contact the patient prior to the visit to remind them of this next visit.

   Week 8 (Visit 4): This study visit will allow collection of eye exam data, vision, eye pressure, and OCT. This visit will last approximately 1 hour. The next study visit (Visit 5) will be scheduled in 4-5 weeks. Someone from the study doctor's office will contact the patient prior to the visit to remind them of this next visit.

   Week 12 (Visit 5): This study visit will allow collection of eye exam data, vision, eye pressure, and OCT. This visit will last approximately 1 hour. The next study visit (Visit 6) will be scheduled in 4-5 weeks. Someone from the study doctor's office will contact the patient prior to the visit to remind them of this next visit.

   Week 16 (Visit 6): This study visit will allow collection of eye exam data, vision, eye pressure, and OCT. This visit will last approximately 1-2 hours. At this visit, the study doctor will determine the need for retreatment with the patient's assigned study treatment regimen. If they do not receive treatment, it is because the initial treatments administered at the baseline (visit 2) are still working and patients will be re-assessed for retreatment at study visit 7. The next study visit (Visit 7) will be scheduled in 4-5 weeks. Someone from the study doctor's office will contact the patient prior to their visit to remind them of this next visit.

   Week 20 (Visit 7): This study visit will allow collection of eye exam data, vision, eye pressure, and OCT. This visit will last approximately 1-2 hours. At this visit, the study doctor will determine the need for retreatment with the patient's assigned study treatment regimen. If they do not receive treatment, it is because the initial treatments administered at the baseline (visit 2) are still working and patients will be re-assessed for retreatment at study visit 8. The next study visit (Visit 8) will be scheduled in 4-5 weeks. Someone from the study doctor's office will contact the patient prior to their visit to remind them of this next visit.

   Week 24 (Visit 8): This study visit will allow collection of eye exam data, vision, eye pressure, and OCT. Additionally; patients will undergo intravenous fluorescein angiogram to assess any changes in your retinal circulation status. This visit will last approximately 2 hours.
3. Post-Randomization Treatment

   Study eyes will be evaluated for retreatment at the week 16 and or week 20 study visits based on BCVA and CST. If an eye experiences a prior treatment-related AE, retreatment is at the discretion of the investigator.

   Retreatments will be deferred if:

   • BCVA letter score is ≥ 84 (20/20 or better) and the SD-OCT CST is < the sex-specific SD-OCT cut-offs below:
   * Zeiss Cirrus: 290 µm in women and 305 µm in men

   Retreatments will be administered if:

   • VA letter score is < 84 (worse than 20/20) and the SD-OCT CST is ≥ the sex-specific SD-OCT cut-offs below:
   * Zeiss Cirrus: 290 µm in women and 305 µm in men If at any time the investigators wish to treat the study eye(s) with a DME treatment that is different from the protocol treatment due to perceived failure or futility communication must be made with the other study investigator.
4. PATIENT WITHDRAWAL & LOSS TO FOLLOW-UP

   A study participant has the right to withdrawal from the study at any time. If a study participant is considering withdrawal from the study, the lead investigator at each respective site should personally discuss with the subject the reasons for discontinuation and every effort should be made to accommodate the patient. Study participants who withdraw will be asked to have a final closeout visit at which time the testing described for the protocol visits will be performed. Study participants who have an AE related to a study treatment or procedure will be asked to continue in follow-up until the AE has resolved or stabilized.
5. Procedures to avoid perception undue influence

The lead investigator and co-investigators for each site will make initial contact in person with the patient. In the informed consent process, the study will be explained to the patients by a study coordinator and all questions of the patients will be answered. A consent form will be given and patients will be given as much time as they need. If needed, the patient may take home the consent form and decide later if they want to participate in the study. Additionally, if the patient cannot read and understand English, a consent form will be provided to them in a language that is understandable to them.

All patients will be assured that the standard of care will be given should the patients choose not to participate in the study. This information is included in the informed consent form and will help patients in their decision.

All patients will be instructed to contact the investigation if they have questions or concerns regarding the study.

7. Statistic Methods

Data will be analyzed using SPSS Statistics software, with the level of statistical significance set at p<0.05.

A single center, 12 month pilot study randomizing 40 DME eyes from 30 subjects 1:1 to BCZ plus adjunctive DEX implant (i.e., BCZ (1.25 mg) at baseline and then monthly when retreatment criteria was met except at months 5 and 10 when DEX implant (0.7 mg) was administered 0.7 mg) or BCZ (1.25 mg monthly) demonstrated similar mean vision gains (+4.9 ± 12.3 ETDRS letters vs. +5.4 ± 10.7 ETDRS letters) but more effective resolution of central subfield thickness (30 ± 100 µm vs. 45 ± 107 µm) with the combination regimen (Maturi RK, 2013; ClinicalTrials.gov Identifier: NCT01309451 http://clinicaltrials.gov/ct2/show/record/NCT01309451). We estimate that a final sample size of at least 20 eyes per study arm is required. Assuming a third of the study eyes may be lost to follow-up we will require enrolment of 30 eyes per study arm.

9. Safety Reporting

All adverse events will be documented and appropriately described. The severity of the adverse event will be coded as mild, moderate, or severe; the association with the intervention will be coded as not related, possibly related or related. The determination of the severity and association will be decided by the principal investigator (PI). The PI for this study will also be acting as the safety monitor, reviewing all adverse events. All serious adverse events that are unexpected and potentially related to the research will be reported in an expedited manner to the research ethical board, the other participating centre and Health Canada.

10. Confidentiality 10.1 Data Confidentiality

All documents relating to the study, including the protocol and data collected during the trial, are the confidential property of the principal investigators.

10.2 Patient Confidentiality

The investigators will preserve the confidentiality of patients participating in the study by identifying them at all times by their study number and will not use patients' names on CRFs or other documentation.

Patients will only be identified on the study database and trial documentation by their assigned study number. All data will be handled in accordance with the Federal Personal Information Protection and Electronic Documents Act (effective January 1, 2004) and all applicable provincial privacy legislation.

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 or 2 diabetic patients
2. Pseudophakic (or phakic without cataract;<1+ nuclear sclerosis) lens status with intact posterior lens capsule and / or Nd:YAG laser capsulotomy that in the investigator's opinion is not likely to permit dislocation of DEX implant into the anterior chamber
3. Center-involved DME > 250 µm
4. Baseline BCVA between 20/40 - 20/320
5. Duration of DME ≤ 9 months
6. Glycosylated haemoglobin (HbA1c) levels ≤ 11%
7. Eyes with intraocular pressure (IOP) ≤ 21 and / or treatment with < 2 topical IOP-lowering medications (eyes with history of previous angle -closure or similar conditions that have been successfully treated with either laser or surgical intervention are allowed as long as the visual fields and optic nerves have been stable for > 1 year prior to study entry and the patient has been and can be safely dilated)
8. Demonstrated incomplete response to 3-6 prior intravitreal anti-VEGFs (AVASTIN®, LUCENTIS®, or EYLEA®; administered every 4 ± 2 weeks over 12-36 weeks (or 3-9 months)); incomplete response is defined herein as a treatment effect resulting in:

   1. < 20% reduction in central subfield thickness (CST) by SD-OCT compared to the baseline first RBZ injection, or
   2. < 5-letter increase in visual acuity compared to the baseline first RBZ injection and/or
   3. the opinion of the treating ophthalmologist additional anti-VEGF monotherapy is not deemed likely to provide further therapeutic benefit
9. If both eyes qualify investigators may enrol bilaterally, with one eye receiving the RBZ plus DEX implant combination regimen and the other receiving the DEX implant monotherapy regimen
10. Written informed patient consent

Exclusion Criteria:

1. Patients with active or suspected ocular or periocular infections including most viral diseases of the cornea and conjunctiva, including active epithelial herpes simplex keratitis (dendritic keratitis), vaccinia, varicella, mycobacterial infections, and fungal diseases.
2. Patients with known hypersensitivity to any components of RBZ or DEX implant
3. Patient has suffered from a stroke or trans-ischemic attack (TIA) in the last 6 months
4. Patients using topical anti-inflammatory medication for the duration of the study
5. Patients with ACIOL (Anterior Chamber Intraocular Lens) and rupture of the posterior lens capsule
6. Prior panretinal or macular laser treatments
7. Previous vitrectomy
8. Any ocular condition that in the opinion of the investigator would not permit improvement of visual acuity with resolution of ME (e.g., foveal atrophy, pigment abnormalities, dense subfoveal hard exudates and/or poor foveal architecture suggestive of photoreceptor loss)
9. Patients with retinal diseases, other than diabetes that can affect ME
10. HbA1c levels > 11%
11. Eyes with a history of advanced glaucoma (optic nerve head change consistent with glaucoma damage and / or glaucomatous visual field loss), uncontrolled ocular hypertension (baseline IOP > 21 mmHg despite use of ≥ 2 topical IOP-lowering medication)
12. Eyes with a history of steroid response (i.e., increase of ≥ 5 mmHg IOP following topical steroid treatment)
13. Eyes with demonstrated response to 3-6 prior monotherapy intravitreal anti-VEGF (i.e., AVASTIN®, LUCENTIS® or EYLEA® administered every 4 ± 2 weeks over 12-36 weeks (or 3-9 months)); response is defined herein as a treatment effect resulting in:

    1. ≥ 20% reduction in CST by SD-OCT from baseline first anti-VEGF injection,
    2. ≥ 5-letter increase in visual acuity since the baseline first anti-VEGF injection and/or,
    3. the opinion of the treating ophthalmologist additional anti-VEGF monotherapy is deemed likely to provide further therapeutic benefit
14. Female patients who are pregnant, breast feeding, or are unable to attend the scheduled follow-up study visits
15. Patients who are unable to attend scheduled follow-up visits throughout the 24-week study
16. Use of systemic steroid, anti-VEGF or pro-VEGF treatment within 4 months prior to enrolment or anticipated use during the study (these drugs are prohibited from use during the study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-11; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Comparison of mean change from baseline ETDRS BCVA letters | From randomization (0) to 24+/- 1 weeks
  Carried out using Area Under the Curve (AUC) analysis

SECONDARY OUTCOMES:
Mean change in Central Subfield Thickness (CST) | From randomization (0) to 24+/- 1 weeks
  Carried out using AUC analysis
Number of re-injections | From randomization (0) to 24+/- 1 weeks
  injections needed in 24 +/- 1 weeks
Re-injection interval | From randomization (0) to 24+/- 1 weeks
  time between injections in 24 +/- 1 weeks
Proportion of eyes with 15- and 10-ETDRS letters gained/lost | From randomization (0) to 24+/- 1 weeks
  percentage of eyes enrolled with 2 and 3 lines gained
Proportion of study eyes with Proliferative Diabetic Retinopathy (PDR) at study completion | From randomization (0) to 24+/- 1 weeks
  percentage of eyes enrolled with neovascularization at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Pradeepa Yoganathan, MD, MSc, Principal Investigator
Locations (2):
- Canada (2):
  - Toronto Retina Institue, Toronto, Ontario
  - North Toronto Eye Care Laser and Eye Specialists, Toronto, Ontario

REFERENCES:
- [Background] Antcliff RJ, Marshall J. The pathogenesis of edema in diabetic maculopathy. Semin Ophthalmol. 1999 Dec;14(4):223-32. doi: 10.3109/08820539909069541. PMID 10758223
- [Background] Antonetti DA, Wolpert EB, DeMaio L, Harhaj NS, Scaduto RC Jr. Hydrocortisone decreases retinal endothelial cell water and solute flux coincident with increased content and decreased phosphorylation of occludin. J Neurochem. 2002 Feb;80(4):667-77. doi: 10.1046/j.0022-3042.2001.00740.x. PMID 11841574
- [Background] Boyer DS, Faber D, Gupta S, Patel SS, Tabandeh H, Li XY, Liu CC, Lou J, Whitcup SM; Ozurdex CHAMPLAIN Study Group. Dexamethasone intravitreal implant for treatment of diabetic macular edema in vitrectomized patients. Retina. 2011 May;31(5):915-23. doi: 10.1097/IAE.0b013e318206d18c. PMID 21487341
- [Background] Boyer DS, Yoon YH, Belfort R Jr, Bandello F, Maturi RK, Augustin AJ, Li XY, Cui H, Hashad Y, Whitcup SM; Ozurdex MEAD Study Group. Three-year, randomized, sham-controlled trial of dexamethasone intravitreal implant in patients with diabetic macular edema. Ophthalmology. 2014 Oct;121(10):1904-14. doi: 10.1016/j.ophtha.2014.04.024. Epub 2014 Jun 4. PMID 24907062
- [Background] Brown DM, Nguyen QD, Marcus DM, Boyer DS, Patel S, Feiner L, Schlottmann PG, Rundle AC, Zhang J, Rubio RG, Adamis AP, Ehrlich JS, Hopkins JJ; RIDE and RISE Research Group. Long-term outcomes of ranibizumab therapy for diabetic macular edema: the 36-month results from two phase III trials: RISE and RIDE. Ophthalmology. 2013 Oct;120(10):2013-22. doi: 10.1016/j.ophtha.2013.02.034. Epub 2013 May 22. PMID 23706949
- [Background] Chang-Lin JE, Attar M, Acheampong AA, Robinson MR, Whitcup SM, Kuppermann BD, Welty D. Pharmacokinetics and pharmacodynamics of a sustained-release dexamethasone intravitreal implant. Invest Ophthalmol Vis Sci. 2011 Jan 5;52(1):80-6. doi: 10.1167/iovs.10-5285. PMID 20702826
- [Background] Cheung N, Mitchell P, Wong TY. Diabetic retinopathy. Lancet. 2010 Jul 10;376(9735):124-36. doi: 10.1016/S0140-6736(09)62124-3. Epub 2010 Jun 26. PMID 20580421
- [Background] Diabetic Retinopathy Clinical Research Network; Elman MJ, Aiello LP, Beck RW, Bressler NM, Bressler SB, Edwards AR, Ferris FL 3rd, Friedman SM, Glassman AR, Miller KM, Scott IU, Stockdale CR, Sun JK. Randomized trial evaluating ranibizumab plus prompt or deferred laser or triamcinolone plus prompt laser for diabetic macular edema. Ophthalmology. 2010 Jun;117(6):1064-1077.e35. doi: 10.1016/j.ophtha.2010.02.031. Epub 2010 Apr 28. PMID 20427088
- [Background] Funatsu H, Noma H, Mimura T, Eguchi S, Hori S. Association of vitreous inflammatory factors with diabetic macular edema. Ophthalmology. 2009 Jan;116(1):73-9. doi: 10.1016/j.ophtha.2008.09.037. PMID 19118698
- [Background] Gillies MC, Sutter FK, Simpson JM, Larsson J, Ali H, Zhu M. Intravitreal triamcinolone for refractory diabetic macular edema: two-year results of a double-masked, placebo-controlled, randomized clinical trial. Ophthalmology. 2006 Sep;113(9):1533-8. doi: 10.1016/j.ophtha.2006.02.065. Epub 2006 Jul 7. PMID 16828501
- [Background] Treatment techniques and clinical guidelines for photocoagulation of diabetic macular edema. Early Treatment Diabetic Retinopathy Study Report Number 2. Early Treatment Diabetic Retinopathy Study Research Group. Ophthalmology. 1987 Jul;94(7):761-74. doi: 10.1016/s0161-6420(87)33527-4. PMID 3658348
- [Background] Haller JA, Bandello F, Belfort R Jr, Blumenkranz MS, Gillies M, Heier J, Loewenstein A, Yoon YH, Jacques ML, Jiao J, Li XY, Whitcup SM; OZURDEX GENEVA Study Group. Randomized, sham-controlled trial of dexamethasone intravitreal implant in patients with macular edema due to retinal vein occlusion. Ophthalmology. 2010 Jun;117(6):1134-1146.e3. doi: 10.1016/j.ophtha.2010.03.032. Epub 2010 Apr 24. PMID 20417567
- [Background] Hooper P, Boucher MC, Colleaux K, Cruess A, Greve M, Lam WC, Shortt S, Tourville E. Contemporary management of diabetic retinopathy in Canada: from guidelines to algorithm guidance. Ophthalmologica. 2014;231(1):2-15. doi: 10.1159/000354548. Epub 2013 Nov 12. PMID 24246998
- [Background] Kiddee W, Trope GE, Sheng L, Beltran-Agullo L, Smith M, Strungaru MH, Baath J, Buys YM. Intraocular pressure monitoring post intravitreal steroids: a systematic review. Surv Ophthalmol. 2013 Jul-Aug;58(4):291-310. doi: 10.1016/j.survophthal.2012.08.003. PMID 23768920
- [Background] Korobelnik JF, Do DV, Schmidt-Erfurth U, Boyer DS, Holz FG, Heier JS, Midena E, Kaiser PK, Terasaki H, Marcus DM, Nguyen QD, Jaffe GJ, Slakter JS, Simader C, Soo Y, Schmelter T, Yancopoulos GD, Stahl N, Vitti R, Berliner AJ, Zeitz O, Metzig C, Brown DM. Intravitreal aflibercept for diabetic macular edema. Ophthalmology. 2014 Nov;121(11):2247-54. doi: 10.1016/j.ophtha.2014.05.006. Epub 2014 Jul 8. PMID 25012934
- [Background] Lazic R, Lukic M, Boras I, Draca N, Vlasic M, Gabric N, Tomic Z. Treatment of anti-vascular endothelial growth factor-resistant diabetic macular edema with dexamethasone intravitreal implant. Retina. 2014 Apr;34(4):719-24. doi: 10.1097/IAE.0b013e3182a48958. PMID 23975006
- [Background] Massin P, Bandello F, Garweg JG, Hansen LL, Harding SP, Larsen M, Mitchell P, Sharp D, Wolf-Schnurrbusch UE, Gekkieva M, Weichselberger A, Wolf S. Safety and efficacy of ranibizumab in diabetic macular edema (RESOLVE Study): a 12-month, randomized, controlled, double-masked, multicenter phase II study. Diabetes Care. 2010 Nov;33(11):2399-405. doi: 10.2337/dc10-0493. PMID 20980427
- [Background] Mitchell P, Bandello F, Schmidt-Erfurth U, Lang GE, Massin P, Schlingemann RO, Sutter F, Simader C, Burian G, Gerstner O, Weichselberger A; RESTORE study group. The RESTORE study: ranibizumab monotherapy or combined with laser versus laser monotherapy for diabetic macular edema. Ophthalmology. 2011 Apr;118(4):615-25. doi: 10.1016/j.ophtha.2011.01.031. PMID 21459215
- [Background] Miyamoto K, Khosrof S, Bursell SE, Rohan R, Murata T, Clermont AC, Aiello LP, Ogura Y, Adamis AP. Prevention of leukostasis and vascular leakage in streptozotocin-induced diabetic retinopathy via intercellular adhesion molecule-1 inhibition. Proc Natl Acad Sci U S A. 1999 Sep 14;96(19):10836-41. doi: 10.1073/pnas.96.19.10836. PMID 10485912
- [Background] Nepomuceno AB, Takaki E, Paes de Almeida FP, Peroni R, Cardillo JA, Siqueira RC, Scott IU, Messias A, Jorge R. A prospective randomized trial of intravitreal bevacizumab versus ranibizumab for the management of diabetic macular edema. Am J Ophthalmol. 2013 Sep;156(3):502-510.e2. doi: 10.1016/j.ajo.2013.04.026. Epub 2013 Jun 21. PMID 23795985
- [Background] Nguyen QD, Brown DM, Marcus DM, Boyer DS, Patel S, Feiner L, Gibson A, Sy J, Rundle AC, Hopkins JJ, Rubio RG, Ehrlich JS; RISE and RIDE Research Group. Ranibizumab for diabetic macular edema: results from 2 phase III randomized trials: RISE and RIDE. Ophthalmology. 2012 Apr;119(4):789-801. doi: 10.1016/j.ophtha.2011.12.039. Epub 2012 Feb 11. PMID 22330964
- [Background] Pacella E, Vestri AR, Muscella R, Carbotti MR, Castellucci M, Coi L, Turchetti P, Pacella F. Preliminary results of an intravitreal dexamethasone implant (Ozurdex(R)) in patients with persistent diabetic macular edema. Clin Ophthalmol. 2013;7:1423-8. doi: 10.2147/OPTH.S48364. Epub 2013 Jul 16. PMID 23901252
- [Background] Tamura H, Miyamoto K, Kiryu J, Miyahara S, Katsuta H, Hirose F, Musashi K, Yoshimura N. Intravitreal injection of corticosteroid attenuates leukostasis and vascular leakage in experimental diabetic retina. Invest Ophthalmol Vis Sci. 2005 Apr;46(4):1440-4. doi: 10.1167/iovs.04-0905. PMID 15790913
- [Background] Wang K, Wang Y, Gao L, Li X, Li M, Guo J. Dexamethasone inhibits leukocyte accumulation and vascular permeability in retina of streptozotocin-induced diabetic rats via reducing vascular endothelial growth factor and intercellular adhesion molecule-1 expression. Biol Pharm Bull. 2008 Aug;31(8):1541-6. doi: 10.1248/bpb.31.1541. PMID 18670086